CLINICAL TRIAL: NCT05382195
Title: Clinical Correlates of Psychiatric Comorbidities in Patients With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Mamdouh Ramadan, resident doctor at Neuropsyiatric department faculty of medicine sohag university, Sohag University
Other Study IDs: Soh-Med-22-05-06
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Patients With Multiple Sclerosis
MeSH Terms: interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: hospital anxiety and depression scale — questionare on patients with multiple sclerosis
  Other Names: multiple sclerosis quality of life 54 intrument

SUMMARY:
Many neuropsychiatric abnormalities associated with multiple sclerosis (MS). These may be broadly divided into 2 categories: disorders of mood, affect,and behavior and abnormalities affecting cognition. With respect to the former, theepidemiology, phenomenology, and theories of etiology are described for the syndromes ofdepression, bipolar disorder, euphoria, pathological laughing and crying, and psychosisattributable to MS.

Finally,treatment pertaining to all these disorders is reviewed, with the observation thattranslational research has been found wanting when it comes to providing algorithms toguide clinicians. Guidelines derived from general psychiatry still largely apply, althoughthey may not always be most effective in patients with neurologic disorders.

The importance of future research addressing this imbalance is emphasized, forneuropsychiatric sequel add significantly to the morbidity associated with MS.(1) The evolution of the neuropsychiatry of multiple sclerosis(MS), with a set sequence of events unfoldingoverthecourseofacenturyormore,providesahistoricalparadigmforotherneurologicdisorders.Accordingtotheparadigm,aclinically astute neurologist, whom posterity will treat kindly,first describes the neurologic (and occasionally, the psycho-logical) signs and symptomsthat cometo define the disorder.

Over succeeding decades, the diagnostic criteria arerefined by further observation supplemented by data fromnew technologies. Mental state changes either pass with littlenoticeoraremissed.Acoupleofgenerationslatercomes belated recognition of prominent abnormalities in mentation-neuropsychiatryredux.

. Invariably, the data reveal major psychiatric problems integral to the disease, and then, with fewexceptions, clinical research stops. Few double-blind,placebo-controlled treatment trials in neuropsychiatry provide an evidence-based approach to treating the newly discernedbehaviouralabnormalities.

ThelifetimeprevalenceofmajordepressioninMS isapproximately 50% (2). A meta-analysis suggests that this is higherthan in other neurologic disorders (3) and, depending on thereferencepoint,is3to10 timestherateinthegeneral population (4). While the basic phenomenology of the MS depressive syndrome overlaps with that found in primarydepression, certain symptoms are more typical, while othersoccur less commonly. Thus, irritability, discouragement, andasenseoffrustration aremorelikelytoaccompanylowmoodthan are feelings of guilt and poor self-esteem (5). It is alsoimportanttorememberthatsymptomssuchasinsomnia,poorappetite,anddifficultieswithconcentrationandmemorymaybe equally attributable to depression or to MS.

Depression is an important reason for so many MS patients'thoughtsofself-harm:suicidalintentoccursinapproximately30% of MS patients and is linked to the presence and severityof depression and social isolation (

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of MS will be established clinically from the history according to revised McDonald's criteria 2010 The following psychiatric disorders ;depression , anxiety fulfilling the diagnostic criteria according to DSM5 as regard therapy, in the out patient clinic of Neuropsychiatry at Sohag university hospital from 1-6-2022 to 1-2-2023

Exclusion Criteria:

* Any patient with the following will be excluded from the study

  1. diagnosis of m.s is not definite
  2. vitally un stable
  3. refused consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
depression in patients with multiple sclerosis | 8 months
  hospital anxiety and depression scale a questionaire of depression from 0 to 21
anxiety in patients with multiple sclerosis | 8 months
  hospital anxiety and depression scale a questionaire of anxiety from 0to 21

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marrie RA, Cohen J, Stuve O, Trojano M, Sorensen PS, Reingold S, Cutter G, Reider N. A systematic review of the incidence and prevalence of comorbidity in multiple sclerosis: overview. Mult Scler. 2015 Mar;21(3):263-81. doi: 10.1177/1352458514564491. Epub 2015 Jan 26. PMID 25623244
- [Background] Wu N, Minden SL, Hoaglin DC, Hadden L, Frankel D. Quality of life in people with multiple sclerosis: data from the Sonya Slifka Longitudinal Multiple Sclerosis Study. J Health Hum Serv Adm. 2007 Winter;30(3):233-67. PMID 18236703
- [Background] Papuc E, Stelmasiak Z. Factors predicting quality of life in a group of Polish subjects with multiple sclerosis: accounting for functional state, socio-demographic and clinical factors. Clin Neurol Neurosurg. 2012 May;114(4):341-6. doi: 10.1016/j.clineuro.2011.11.012. Epub 2011 Dec 1. PMID 22137087
- [Background] Feinstein A. The neuropsychiatry of multiple sclerosis. Can J Psychiatry. 2004 Mar;49(3):157-63. doi: 10.1177/070674370404900302. PMID 15101497